CLINICAL TRIAL: NCT02968745
Title: Occupational Performance Problems Frequently Reported by Individuals With Rheumatoid Arthritis
Brief Title: Occupational Performance Problems in Individuals With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Júnia Amorim Andrade, PHD Júnia Amorim Andrade, Federal University of Minas Gerais
Other Study IDs: UFMG ETIC 024/09
Record Dates: First submitted 2016-11-13; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: RheumatoId Arthritis
Keywords: Rheumatoid arthritis; human activity; Canadian Occupational Performance Measure
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational study — Canadian Occupational Performance Measure (COPM) was applied to identify the main occupational performance problems

SUMMARY:
Aim: To identify the main occupational performance problems reported by individuals with rheumatoid arthritis and the relationship between these activities with work status of participants . Methods: the investigators conducted a cross-sectional study with 81 patients with RA. Individuals were interviewed the Canadian Occupational Performance Measure. Data was described in frequencies and percentages, and the Pearson's chi-square test was used to determine the asymptotic association between the occupational performance problems with work.

DETAILED DESCRIPTION:
For this cross-sectional study, 81 patients were recruited by convenience at the Clinical Hospital (HC) of the Universidade Federal de Minas Gerais (UFMG), in Brazil.

COPM was applied to identify the main occupational performance problems reported by participants. The COPM is an individual measure of self-awareness about the problems faced when carrying out the activities. It identifies problems in the areas of self-care, productivity, and leisure, and measure the individual's performance and satisfaction regarding these activities

ELIGIBILITY:
Inclusion Criteria:

* over 46 years old;
* diagnosed with RA by rheumatologist (American College of Rheumatology);
* mental competency as assessed with the Mental State Mini-Examination;
* possessed the skills to understand the instructions study.

Exclusion Criteria

* had undergone surgery in the upper limbs.

Ages: 46 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For this cross-sectional study, 81 patients treated between 2009 and August 2010 in clinical Hospital, at the Universidade Federal de Minas Gerais (UFMG) in Brazil werw recruited by convenience sampling
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | June 2009 to August 2010
  The COPM protocol is divided into three areas: self-care, productivity, and leisure. Patients define important activities and classify them with a score of one to 10 (a score of one indicated no importance and a score of 10 indicated extreme importance),

IPD SHARING:
Plan to Share IPD: No
Not plan to Share IPD